CLINICAL TRIAL: NCT03376373
Title: Neurotherapy to Promote Emotion Recognition in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, John Richey, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH100268
Record Dates: First submitted 2016-12-18; First posted 2017-12-18 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: independent evaluators are masked to condition assignment
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (Experimental): Neurofeedback for FER
  Interventions: Behavioral: neurofeedback
- control (No Intervention): waiting list

INTERVENTIONS:
Behavioral: neurofeedback — real-time feedback on accuracy of emotion recognition
  Arms: active

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder, more prevalent than previously thought and heterogeneous in expression, though uniformly characterized by severe social disability. The social disability that defines ASD pervades other areas of adaptive behavior, is predictive of secondary mental health problems, and adversely affects long-term outcome. Although ASD is a chronic condition, there has been little research on interventions for adults with ASD. This study proposes to first establish the neural plasticity of specific brain mechanisms underlying difficulties with facial emotion recognition, a core deficit believed to be pivotal in the behavioral expression of ASD-social disability. The investigators will then develop a novel, computer-based intervention using real-time feedback, to the user, to ameliorate emotion recognition deficits.

DETAILED DESCRIPTION:
Individuals with autism spectrum disorder (ASD) are known to have difficulty in the recognition of facial emotion. Such deficits in facial emotion recognition (FER) are thought to cause or exacerbate social disability in ASD by preventing 1) accurate detection of social/emotional information conveyed through the face and, subsequently 2) the deployment of emotionally appropriate responses. Consistent with this model, FER deficits are correlated with social disability in ASD and confer morbidity above and beyond core symptoms.

The long-term goal is to understand how FER networks can be manipulated for therapeutic and preventative purposes. In this trial, investigators are testing the feasibility of an intervention that capitalizes on our previously developed brain-computer interface (BCI) to promote FER in a mixed virtual reality world. The new "FER Assistant" tool (deployed on a tablet - iPad) is intended to aid users in detecting emotions and intents of 'avatars' inhabiting a virtual world, and will provide users with a highly realistic testbed for practicing FER skills in concert with BCI.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ASD

Exclusion Criteria:

* No severe psychopathology which warrants other immediate treatment

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
facial emotion recognition (RMET) | 5 weeks
  Change in facial emotion recognition 5 weeks after baseline appointment

CONTACTS AND LOCATIONS:
Overall Officials: Richey, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Child Study Center, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No